CLINICAL TRIAL: NCT03063840
Title: To Evaluate the Safety and Efficacy of Microwave Ablation for the Treatment of Malignant
Brief Title: Microwave Ablation for the Treatment of Malignant Liver Tumors Closed to Intrahepatic Vessels
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NO participants enrolled
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201603095DIPD
Record Dates: First submitted 2017-01-04; First posted 2017-02-24 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Liver Cancer
Keywords: hepatocellular carcinoma; microwave ablation; liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Microwave ablation (MWA) (Experimental): Microwave ablation (MWA)
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Microwave ablation (MWA): Emprint Microwave Ablation system with 2.45 GHz microwave generator

SUMMARY:
Liver cancer including primary hepatocellular carcinoma (HCC) and metastatic liver cancers is one the most common malignancies in the world. Over 10000 new cases per year are diagnosed in Taiwan. Despite the many treatment options, the prognosis of HCC remains dismal. More than 8000 people died of this cancer every year in Taiwan. A majority (70% to 85%) of patients present with advanced or unresectable disease. In contrast, small liver cancers can be cured with an appreciable frequency. Five-year disease-free survival exceeding 50% has been reported for surgical resection, and for the inoperable patients who do not have vascular invasion or extrahepatic spread. Radiofrequency ablation (RFA) is recommended as an alternative curative therapy. However, the main drawback of RFA is its limitation to tumor size and location. The tumors larger than 5 cm in diameter or located adjacent to vessels, could not be ablated completely sometimes. Microwave ablation (MWA) can ablate tumor by higher temperature than RFA, so is supposed not to be diminished by adjacent vessels.

DETAILED DESCRIPTION:
Several pre-clinical studies have already demonstrated microwave ablation (MWA) is a safe and effective treatment for live cancers. The system (Emprint Microwave Ablation system) with 2.45 GHz microwave generator the investigators will use has been approved as safe by the European Union (EU) in 2009 and received Food and Drug Administration (FDA) approval in 2014. However, there are still few experiences in using MWA for tumor ablation in Taiwan. In this study, we will perform MWA for 40 inoperable patients with liver cancers adjacent to vessels who are suitable to receive radiofrequency ablation (RFA) in our hospital. The investigators will evaluate the potential side effect and ablate effect of tumors by abdominal computed tomography (CT) or magnetic resonance imaging (MRI), and the investigators will also follow-up this patients for 1 years to evaluate the overall survival and local recurrence rate. The investigators will appraisal the clinical feasibility and advantage of the system by this study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Unsuitable for surgical resection but local ablation is indicated, however, the distance between tumour and vessels is smaller than 1 cm.
2. Have at least one, but less than or equal to 3 tumors.
3. Each tumor must be ≤ 5 cm in diameter.
4. Child-Pugh class A-B.
5. Eastern Cooperative Oncology Group (ECOG) score of 0-1.
6. American Society of Anaesthesiologists (ASA) score ≤ 3.
7. Adequate bone marrow and liver function (1). Platelet count ≥ 100 K/Μl(2). Total bilirubin ≦ 2 mg/dL(3). alanine transaminase (ALT) and aspartate transaminase (AST) < 5 x upper limit of normal (4). prothrombin time (PT)- international normalized ratio (INR) ≦ 2.0.
8. The disease status is not suitable to receive transarterial chemoembolization or other standard treatment.
9. Prior Informed Consent Form.
10. Life expectancy of at least 3 months.

Exclusion Criteria:

Patients presenting with any of the following will not be enrolled into this study:

1. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception.
2. Received treatment with an investigational agent/ procedure within 30 days prior to microwave ablation.
3. Patients who cannot tolerate radiofrequency ablation (RFA) procedure.
4. Known history of human immunodeficiency virus (HIV) infection.
5. Concurrent extrahepatic cancer.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
tumor evaluation | 1 month after treatment
  Tumor response will be evaluated by abdominal computed tomography (CT) or magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) evaluation | up to two years
  Complete an Eastern Cooperative Oncology Group (ECOG) evaluation
Clinical laboratory assessment | up to two years
  Collect blood sample for hematology evaluation
Conduct computed tomography (CT) or magnetic resonance imaging (MRI) scans for tumour response evaluation | up to two years
  Subjects will still be followed-up in the event of disease progression in order to document local recurrence.
Review concomitant medications | up to two years
  Use of medications will be reviewed and recorded
Assess for presence of adverse events | up to two years
  An adverse event assessment will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No